CLINICAL TRIAL: NCT06211179
Title: An Open-label, Randomized, Single-dose, Three-way Crossover Study to Assess the Relative Bioavailability of 5 mg Mavacamten Opened Capsule Administered Via Nasogastric Tube Compared to 5 mg Mavacamten Intact Capsule in Healthy Participants
Brief Title: A Study to Assess the Relative Bioavailability of 5 mg Mavacamten Opened Capsule Administered Via Nasogastric Tube Compared to Intact Oral 5 mg Mavacamten in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CV027-1070
Record Dates: First submitted 2023-12-18; First posted 2024-01-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sequence ABC (Experimental)
  Interventions: Drug: Treatment A: Mavacamten intact oral capsule; Drug: Treatment B: Mavacamten open capsule in suspension; Drug: Treatment C: Mavacamten open capsule in suspension administered via nasogastric tube (NGT)
- Sequence BCA (Experimental)
  Interventions: Drug: Treatment A: Mavacamten intact oral capsule; Drug: Treatment B: Mavacamten open capsule in suspension; Drug: Treatment C: Mavacamten open capsule in suspension administered via nasogastric tube (NGT)
- Sequence CAB (Experimental)
  Interventions: Drug: Treatment A: Mavacamten intact oral capsule; Drug: Treatment B: Mavacamten open capsule in suspension; Drug: Treatment C: Mavacamten open capsule in suspension administered via nasogastric tube (NGT)

INTERVENTIONS:
Drug: Treatment A: Mavacamten intact oral capsule — Specified dose on specified days
Drug: Treatment B: Mavacamten open capsule in suspension — Specified dose on specified days
Drug: Treatment C: Mavacamten open capsule in suspension administered via nasogastric tube (NGT) — Specified dose on specified days

SUMMARY:
The purpose of this study to assess the relative bioavailability of 5 mg Mavacamten opened capsule administered via nasogastric tube compared to intact oral 5 mg Mavacamten in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a body mass index between 18 and 32 kg/m2.
* Participants must be healthy, as determined by physical examination, vital signs, ECGs, and clinical laboratory assessments.
* Participants must be willing and able to adhere to the prohibitions and restrictions specified in the protocol.

Exclusion Criteria:

* Participants must not have any significant acute or chronic medical illness.
* Participants must not have any current or recent (within 3 months of study intervention administration) gastrointestinal disease including, but not limited to, bowel obstruction or perforation, gastrointestinal ulcers, esophageal varices, Crohn's disease, diverticulitis, irritable bowel syndrome, ileus, a gastrointestinal tract that is not anatomically intact, dyspepsia, constipation, diarrhea, or vomiting.
* Participants must not be intolerant or allergic to lidocaine or cetacaine or any type of topical anesthetic.

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to 37 days
Area under the concentration-time curve from time 0 to the last quantifiable time point (AUC[0-T]) | Up to 37 days
Area under the concentration-time curve from time 0 to 72 hours (AUC[0-72]) | Up to 37 days
Area under the concentration-time curve from time 0 to infinite time (AUC[0-INF]) | Up to 37 days

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) | Up to 37 days
Terminal half-life (T-HALF) | Up to 37 days
Apparent clearance (CLT/F) | Up to 37 days
Apparent volume of distribution (Vz/F) | Up to 37 days
Number of participants with adverse events (AEs) | Up to 37 days
Number of participants with serious adverse events (SAEs) | Up to 37 days
Number of participants with vital sign abnormalities | Up to 37 days
Number of participants with electrocardiogram (ECG) findings | Up to 37 days
Number of participants with physical examination findings | Up to 37 days
Number of participants with abnormalities in clinical laboratory evaluations | Up to 37 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-andresearch/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com